CLINICAL TRIAL: NCT03834584
Title: A Phase 1 Study of AG-636 in the Treatment of Subjects With Advanced Lymphoma
Brief Title: A Study of AG-636 in the Treatment of Subjects With Advanced Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to sponsor decision.
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AG636-C-001
Record Dates: First submitted 2019-02-06; First posted 2019-02-08 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Lymphoma
Keywords: Lymphoma; DHODH; Hodgkins Lymphoma; Non-Hodgkins Lymphoma; T-Cell Lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, Non-Hodgkin; Lymphoma, T-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AG-636 (Experimental): AG-636 dosed orally.
  Interventions: Drug: AG-636

INTERVENTIONS:
Drug: AG-636 — AG-636 will be administered orally intermittently in 28-day cycles.

SUMMARY:
This study will evaluate the safety, pharmacokinetics, pharmacodynamics, and clinical activity of AG-636, an oral Dihydroorotate Dehydrogenase (DHODH) inhibitor, in subjects with advanced lymphoma.

DETAILED DESCRIPTION:
The purpose of this Phase 1, multicenter, open-label study is to determine the maximum tolerated dose (MTD) of AG-636 and characterize its dose-limiting toxicities (DLTs) when given by mouth to subjects with advanced lymphoma that is refractory to standard treatment. During the dose escalation part of the study successive cohorts of subjects will be treated with increasing doses of AG-636 in order to determine its maximum tolerated dose (MTD). Subsequently, in the dose expansion part of the study, additional subjects will be treated at the MTD in order to confirm that dose's safety, tolerability, PK and PD, and to provide an opportunity to detect anti-lymphoma activity. The dose expansion part of the study will support the selection of a dose for future clinical studies (a recommended Phase 2 dose [RP2D]).

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥18 years of age.
2. Have a pathologically confirmed diagnosis of a non-Hodgkin or Hodgkin lymphoma that has progressed in spite of prior treatment, and for whom additional effective (curative or life-prolonging) standard therapy is not available. The lymphomas included in this study must fall within one of the following 2017 World Health Organization categories:

   1. Mature B-cell neoplasms (excluding plasma cell neoplasms, heavy chain disease, and primary central nervous system [CNS] lymphoma)
   2. Mature T- and NK-cell neoplasms
   3. Hodgkin lymphomas
   4. Immunodeficiency-associated lymphoproliferative disorders
3. In the case of subjects who have lymphoma for which high-dose chemotherapy and autologous stem cell transplantation (HD-ASCT) is considered a standard curative therapy, eligibility for this study requires that the subject's disease has relapsed after HD-ASCT, that the subject is not eligible for HD-ASCT, or that the subject has refused HD-ASCT.
4. Have disease that can be clinically evaluated for improvement or progression. In the dose expansion phase of the study, subjects must have disease that is measurable (as defined by either the Lugano criteria for lymphoma or the 2011 ISCL/USCLC/EORTC criteria for MF/SS).
5. Have an Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
6. Have an absolute neutrophil count (ANC) ≥1,000/uL.
7. Have a platelet count ≥75,000/uL.
8. Have a serum total bilirubin level ≤1.5×ULN (upper limit of normal) in the absence of Gilbert syndrome. Subjects with Gilbert syndrome must have a serum total bilirubin level ≤1.5× their baseline value.
9. Have alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels ≤3.0×ULN, unless due to underlying hematologic malignancy. If ALT/AST elevations are determined to be due to involvement by the underlying hematologic malignancy, subjects must have ALT/AST levels <5.0× the ULN.(Note: There are no specific requirements for alkaline phosphatase [ALP].)
10. Have a creatinine clearance (CrCl) ≥ 30 mL/min (either measured or estimated by the Cockcroft-Gault formula). (Cockcroft-Gault formula for estimated creatinine clearance [eCrCl]: eCrCl = [140 - Age] × Weight [kg] × [0.85 if Female] / [72 × serum creatinine (mg/dL)]).
11. Be fully recovered from major surgery and from the acute toxic effects of prior chemotherapy and radiotherapy. Residual chronic toxicities of prior therapy, eg, alopecia, Grade ≤2 peripheral neuropathy, are allowed.
12. If female with reproductive potential, must have a negative serum pregnancy test prior to the start of study therapy. Females of reproductive potential, as well as fertile men and their female partners of reproductive potential, must agree to use 2 effective forms of contraception.
13. Able to understand and have provided written informed consent.

Exclusion Criteria:

1. Have a primary central nervous system (CNS) lymphoma.
2. Have lymphomatous involvement of the CNS that is symptomatic or requires therapy. However, subjects who have completed treatment for lymphoma involving the CNS and have no further evidence of disease in the CNS may be enrolled in this study.
3. Have lymphoma that requires immediate cytoreductive therapy.
4. Have low-grade lymphoma that does not meet conventional criteria for requiring treatment.
5. Have impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of AG-636, including any unresolved nausea, vomiting, or diarrhea that is National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade >1.
6. Are unable to abstain from food or liquids other than water for 2 hours before and 2 hours after each dose of AG-636.
7. Have an active infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.
8. Have an active infection (bacterial, viral, or fungal) that cannot be controlled with treatment.
9. Have had significant active cardiac disease within 6 months prior to the start of study treatment, including any of the following:

   1. New York Heart Association (NYHA) class III or IV congestive heart failure.
   2. Acute myocardial infarction or angina pectoris.
   3. Stroke.
   4. Uncontrolled cardiac arrhythmia (subjects with rate-controlled atrial fibrillation are not excluded).
10. Have a heart rate-corrected QT interval using Fridericia's method (QTcF) >470 msec. Patients with bundle branch block and a QTcF >470 msec should be discussed with the Medical Monitor for potential inclusion.
11. Have any other concurrent severe and/or uncontrolled concomitant medical condition that could compromise participation in the study (eg, clinically significant pulmonary disease, clinically significant neurologic disorder).
12. Have received any systemic anticancer treatment or radiotherapy less than 2 weeks before the first dose of AG-636.
13. Have received radioimmunotherapy less than 6 weeks before the first dose of AG-636.
14. Have received treatment with an investigational small molecule <2 weeks before the first dose of AG-636.
15. Are taking medications that are sensitive substrates of CYP2C8, and that cannot be discontinued prior to starting treatment with AG-636.
16. Are taking medications that are sensitive substrates of either P-glycoprotein (P-gp) or breast cancer resistance protein (BCRP), and that cannot be discontinued prior to starting treatment with AG-636.
17. Are pregnant or breastfeeding.
18. Have any other medical or psychological condition deemed by the Investigator to be likely to interfere with the subject's ability to give informed consent or participate in the study.
19. Have concurrent malignancy other than lymphoma; subjects must have been free of other malignancies for ≥1 year before the start of study treatment. However, subjects with the following history/concurrent conditions are allowed:

    1. Basal or squamous cell carcinoma of the skin
    2. Carcinoma in situ of the cervix
    3. Carcinoma in situ of the breast
    4. Incidental histologic finding of prostate cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2020-06-17 (Actual); Study Completion 2020-06-17 (Actual)

PRIMARY OUTCOMES:
The frequency of dose limiting toxicities (DLTs) associated with AG-636 administration during the first cycle (first 28 days) of treatment. | Up to 28 days, on average

SECONDARY OUTCOMES:
Characterize the Safety and Tolerability of AG-636 (number of treatment-related Adverse Events and Serious Adverse Events) | Up to 24 weeks, on average
  As determined by the number of treatment-related Adverse Events and Serious Adverse Events
Characterize the Pharmacodynamics of AG-636 | Up to 24 weeks, on average
  Measured by changes from baseline in circulating upstream metabolites
Pharmacokinetics of AG-636 in plasma | Up to 24 weeks, on average
  Determined by the plasma concentration versus time profile of AG-636
Clinical activity of AG-636 in Lymphoma | Up to 24 weeks, on average
  Assessed by either the Lugano criteria for lymphoma or the 2011 International Society for Cutaneous Lymphomas (ISCL)/United States Cutaneous Lymphoma Consortium (USCLC)/ European Organization for Research and Treatment of Cancer (EORTC) criteria for mycosis fungoides (MF)/Sézary syndrome (SS)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Yale Cancer Center, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No